CLINICAL TRIAL: NCT06325956
Title: Prediction of Immune Status on the Efficacy of Metformin in the Treatment of Polycystic Ovary Syndrome
Brief Title: PCOS Immune Function Predicts Metformin Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Prof., Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immune status and metformin
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome; Metformin; Immune Function
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin therapy (Experimental): Metformin intervention, 1000mg daily for the first week, 1500mg daily starting in the second week until six months of treatment.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Take metformin for six months.
  Other Names: Metformin therapy

SUMMARY:
In this study, the investigators will include PCOS patients who meet the trial criteria, introduce participants to the content of this study, and invite participants to participate. The immune function of peripheral blood samples of PCOS patients was detected by flow cytometry. Participants were further treated with metformin for 6 months and followed up after the intervention. The objective of this study was to investigate immune markers related to the efficacy of metformin in PCOS patients and to predict the efficacy of metformin in PCOS patients using immune function.

DETAILED DESCRIPTION:
In this study, peripheral blood samples of PCOS patients were collected before and after intervention. Flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and fluorescently labeled antibodies in human peripheral blood, and the unlabeled cells were dissolved. The number and percentage of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years
* Diagnosis of PCOS with the Rotterdam diagnosis criteria (2003)

Exclusion Criteria:

* Pregnant women;
* Hyperthyroidism or hypothyroidism
* Severe liver and kidney function injury
* Cancer patients;
* Associated with severe infection, severe anemia, neutropenia and other blood system diseases;
* Have type 1 diabetes, single-gene mutated diabetes or other secondary diabetes;
* Patients with mental illness or intellectual disability;
* Have taken drugs for PCOS treatment in the last three months;
* Have a long history of taking hormone therapy;
* Currently or recently participating in another clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry. | Samples to be collected once per participant within 7 days of enrollment.
  Flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and the fluorescently labeled antibody in human peripheral blood, and the unlabeled cells were dissolved.
The percentage of cell groups expressing different markers were counted by the fluorescence detection system on flow cytometry. | Samples to be collected once per participant within 7 days of enrollment.
  Flow cytometry was used to detect the antigenic antibody reaction between the surface differentiation antigen of lymphocyte membrane and the fluorescently labeled antibody in human peripheral blood, and the unlabeled cells were dissolved.

SECONDARY OUTCOMES:
Homeostasis model assessment of insulin resistance | Within 7 days of enrollment.
  insulin resistance index
body mass index | Within 7 days of enrollment.
  body mass index (kg/m2)
menstrual frequency | Within 7 days of enrollment.
  number of menstruation in a year
fasting glucose | Within 7 days of enrollment.
  fasting glucose (mmol/L)
fasting insulin | Within 7 days of enrollment.
  fasting insulin (mmol/L)
Total cholesterol | Within 7 days of enrollment.
  Total cholesterol (mmol/L)
Triglycerides | Within 7 days of enrollment.
  Triglycerides (mmol/L)
HDL-c | Within 7 days of enrollment.
  HDL-c (mmol/L)
LDL-c | Within 7 days of enrollment.
  LDL-c (mmol/L)
total testosterone | Within 7 days of enrollment.
  total testosterone (nmol/L)
free testosterone | Within 7 days of enrollment.
  free testosterone (nmol/L)
Sex hormone-binding globulin | Within 7 days of enrollment.
  Sex hormone-binding globulin (nmol/L)
Androstenedione | Within 7 days of enrollment.
  Androstenedione (ng/ml)
Dehydroepiandrosterone | Within 7 days of enrollment.
  Dehydroepiandrosterone (ug/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Manna Zhang, doctor, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No